CLINICAL TRIAL: NCT04557059
Title: A Randomized, Controlled, Multicenter, Open-label Study to Investigate the Efficacy and Safety of Adding Apalutamide to Radiotherapy and LHRH Agonist in High-Risk Patients With Hormone-Sensitive Prostate Cancer, Assessed by PSMA-PET With an Observational Cohort
Brief Title: A Study of Adding Apalutamide to Radiotherapy and LHRH Agonist in High-Risk Patients With Hormone-Sensitive Prostate Cancer
Acronym: PRIMORDIUM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108705; 56021927PCR3015 (Other: Janssen Research & Development, LLC); 2019-002957-46 (EudraCT Number); 2023-505852-23-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-09-17; First posted 2020-09-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interventional Cohort (Group 1): RT+ LHRHa (Active Comparator): Participants will receive radiotherapy (RT) which is defined as prostate-bed plus pelvic lymph node salvage external-beam radiotherapy with or without optional stereotactic body radiation therapy (SBRT), along with a luteinizing hormone-releasing hormone agonist (LHRHa) as a 3-monthly depot preparation within 3 days after randomization and the end of Week 12, or as a 6-monthly depot preparation within 3 days after randomization.
  Interventions: Radiation: Radiotherapy; Drug: LHRHa
- Interventional Cohort (Group 2): RT+LHRHa + Apalutamide (Experimental): Participants will receive prostate-bed plus pelvic lymph node salvage external-beam radiotherapy (RT) with or without optional stereotactic body radiation therapy (SBRT), along with a LHRHa as a 3-monthly depot preparation within 3 days after randomization and the end of Week 12, or as a 6-monthly depot preparation within 3 days after randomization. Participants will also receive 240 milligram (mg) of apalutamide starting within 3 days after randomization as film-coated tablets, to be swallowed whole and together once daily with or without food, for a period of 180 Days.
  Interventions: Radiation: Radiotherapy; Drug: LHRHa; Drug: Apalutamide
- Observational Cohort(Group3) PSMA-PET Negative Participants (No Intervention): Enrollment into this cohort will be stopped further. Participants who were PSMA-PET-negative at screening and were already enrolled in the Observational Cohort will continue in this cohort. Data collected in the course of routine clinical practice during this period will include clinical evaluations, disease progression, therapies administered as per standard-of-care at the study-sites and survival status. For Observational Cohort, information will be entered into the electronic case report form (eCRF) from the medical records at least twice a year. The use of any medicinal product(s) for the treatment and management of participants will be at discretion of the treating physician.

INTERVENTIONS:
Radiation: Radiotherapy — Participants will receive radiotherapy (RT) with or without optional stereotactic body radiation therapy (SBRT), which will start within 4 weeks after randomization.
  Arms: Interventional Cohort (Group 1): RT+ LHRHa; Interventional Cohort (Group 2): RT+LHRHa + Apalutamide
Drug: LHRHa — Participants will be administered with LHRHa (example, leuprolide, goserelin, triptorelin acetate) as a 3-monthly depot preparation within 3 days after randomization and the end of Week 12 or as a 6-monthly depot preparation within 3 days after randomization.
  Arms: Interventional Cohort (Group 1): RT+ LHRHa; Interventional Cohort (Group 2): RT+LHRHa + Apalutamide
Drug: Apalutamide — Participants will receive therapeutic dose of apalutamide 240 mg once daily for 180 Days.
  Other Names: JNJ-56021927
  Arms: Interventional Cohort (Group 2): RT+LHRHa + Apalutamide

SUMMARY:
The main purpose of this study is to determine if the addition of apalutamide to radiotherapy (RT) plus luteinizing hormone-releasing hormone agonist (LHRHa) delays metastatic progression as assessed by prostate specific membrane antigen-positron emission tomography (PSMA-PET) or death compared with RT plus LHRHa alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Previously treated with radical prostatectomy with or without lymph node dissection and either: a) for biochemical recurrence after radical prostatectomy (RP): any post-operative prostate-specific antigen (PSA) measurement of less than (<) 0.1 nanogram/milliliter (ng/mL) within 12 months after RP and without any PSA greater than and equal to (>=) 0.1 ng/mL within the 4 to 8-week period after RP or b) for persistent PSA after RP: PSA >=0.1 ng/mL within the 4 to 8-week period after RP, confirmed by additional measurement at least 3 weeks later
* Be able to swallow whole the study drug tablets or follow the instructions for admixing with apple sauce
* Results of the Prostate specific membrane antigen-positron emission tomography (PSMA-PET) at screening as determined by blinded independent, central review (BICR), must be: PSMA-PET-negative for any prostate cancer lesions (that is, no loco-regional lesion and no distant lesions); or PSMA-PET-positive for at least one loco-regional (pelvic) lesion without distant extra-pelvic lesion; or PSMA PET- positive for at least one loco--regional (pelvic) lesion with extra-pelvic lesion(s).
* High risk of developing metastasis defined as; a) for biochemical recurrence after RP: pathological Gleason score greater than or equal to (>=) 8 evaluated from prostate tissue specimen at radical prostatectomy, or prostate-specific antigen doubling time (PSADT) less than or equal to (<=) 12 months at the time of screening; b) for persistent PSA after RP: pathological Gleason score >=8, evaluated from prostate tissue specimen at radical prostatectomy
* Participants with evidence of distant metastasis on screening PSMA-PET scan must have no evidence of prostate cancer metastases on screening CT/MRI of the chest/abdomen/pelvis, Technetium 99m [99mTc] whole-body bone scan. Participants with a single bone lesion on 99mTc whole-body bone scan should have confirmatory imaging by CT or MRI; if the confirmatory scan confirms the bone lesion, the participant should be excluded from the study. Conventional images (99mTc-bone scan and CT/MRI) from the screening will be evaluated locally before randomization
* Eastern Cooperative Oncology Group Performance Status Grade 0 or 1

Exclusion Criteria:

* History of pelvic radiation for malignancy
* Previous treatment with androgen deprivation therapy (ADT) for prostate cancer
* Previously treated for biochemical recurrence (BCR) or persistent PSA after RP (previous surgical treatment of one or more loco-regional lesions is allowed)
* Prior treatment with a CYP17 inhibitor (example, oral ketoconazole, orteronel, abiraterone acetate, galeterone) or any androgen receptor (AR) antagonist including bicalutamide, flutamide, nilutamide, apalutamide, enzalutamide or darolutamide and any other medications that may lower androgen levels (estrogens, progestins, aminoglutethimide, etc.), including bilateral orchiectomy
* Known or suspected contraindications or hypersensitivity to apalutamide, Luteinizing Hormone-Releasing Hormone (LHRH) agonist or any of the components of the formulations
* Prior chemotherapy for prostate cancer
* Any evidence of prostate cancer metastasis on computed tomography/magnetic resonance imaging (CT/MRI) of the chest/abdomen/pelvis or 99mTc whole-body bone scan, at any time prior to screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 694 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2029-08-27 (Estimated); Study Completion 2029-08-27 (Estimated)

PRIMARY OUTCOMES:
Prostate specific Membrane Antigen-Positron Emission Tomography (PSMA-PET) Metastatic Progression-free Survival (ppMPFS) | Up to 9 years
  ppMPFS is defined as the appearance of at least one new PSMA-PET-positive distant lesion compared with the previous scan as assessed by blinded independent central review (BICR) or death.

SECONDARY OUTCOMES:
Time to Prostate-Specific Antigen (PSA) Progression | Up to 9 years
  Time to PSA progression is defined as the time from randomization to the date of first documentation of PSA progression. PSA progression is defined as a PSA concentration above the nadir of more than 0.5 nanogram per milliliter (ng/mL), confirmed by additional measurement at least 3 Weeks later.
PSA Response Rate | Up to 9 years
  PSA response rate is defined as the percentage of participants with a PSA decrease of >= 50 percent (%), >= 90% or undetectable from baseline.
PSA Levels at Week 26 | Week 26
  PSA levels at week 26 will be reported.
Time to Loco-Regional Progression by PSMA-PET | Up to 9 years
  Time to loco-regional progression by PSMA-PET as assessed by blinded independent central review (BCIR) is defined as the time from randomization to the date of the first occurrence of PSMA-PET loco-regional progression. Criteria for PSMA-PET loco-regional progression: Appearance of at least one new PSMA-PET-positive loco-regional lesion compared with the previous scan.
Overall Survival | Up to 9 years
  Overall survival is defined as the time from randomization to date of death from any cause.
Prostate Cancer-Specific Survival | Up to 9 years
  Prostate cancer-specific survival is defined as the time from randomization to date of death due to prostate cancer.
Number of Participants With Adverse Event (AE) and Serious Adverse Events (SAEs) | Up to 9 years
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. An SAE is any AE that results in: death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and is a suspected transmission of any infectious agent via a medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (141):
- United States (13):
  - Arizona Urology Specialists, Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Colorado Clinical Research, Lakewood, Colorado
  - Urological Research Network, Hialeah, Florida
  - First Urology, PSC, Jeffersonville, Indiana
  - Michigan Institute of Urology, Troy, Michigan
  - Associated Medical Professionals of Ny, Syracuse, New York
  - The Urology Group, Cincinnati, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Urology Austin, Austin, Texas
  - Houston Metro Urology, Houston, Texas
  - Spokane Urology, Spokane, Washington
- Australia (8):
  - Bundaberg Hospital, Bundaberg
  - Hervey Bay Hospital, Bundaberg
  - Epworth Healthcare, East Melbourne
  - St Vincent's Hospital - Melbourne, Fitzroy
  - Genesis Care Hurstville, Hurstville
  - Macquarie University Hospital, North Ryde
  - Calvary Mater Newcastle, Waratah
  - GenesisCare Wembley, Wembley
- Austria (3):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Universitaetsklinikum Salzburg Landeskrankenhaus, Salzburg
  - Medizinische Universitaet Wien, Vienna
- Belgium (4):
  - ZAS Augustinus, Antwerp
  - A.Z. Sint Jan, Bruges
  - UZ Gent, Ghent
  - Az Groeninge, Kortrijk
- Brazil (11):
  - Empresa Brasileira de Servicos Hospitalares - EBSERH - Hospital das Clinicas da UFMG, Belo Horizonte
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Hospital Sao Rafael, Salvador
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital Sao Camilo Unidade Vila Mariana, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- Czechia (4):
  - Fakultni nemocnice Plzen, Urologicka klinika, Pilsen
  - Urocentrum Praha, Prague
  - Urologicka klinika 1 LF UK a VFN, Prague
  - Fakultni nemocnice v Motole, Prague
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen N
  - Gentofte Herlev Hospital, Herlev
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
  - Vaasa Central Hospital, Vaasa
- Germany (6):
  - Vivantes Klinikum Am Urban, Berlin
  - Städtisches Klinikum Braunschweig gGmbH - Standort Salzdahlumer, Braunschweig
  - Universitatsklinikum Carl Gustav Carcus Dresden, Dresden
  - Universitatsklinikum Essen, Essen
  - Klinikum rechts der Isar - der Technischen Universität München, München
  - Universitaetsklinikum Muenster, Münster
- Hungary (7):
  - Péterfy Sándor utcai Kórház, Budapest
  - Budapesti Bajcsy Zsilinszky Korhaz es Rendelointezet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Eszak Budai Szent Janos Centrumkorhaz, Budapest
  - Budapesti Uzsoki Utcai Korhaz, Budapest
  - Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- Italy (6):
  - Radioterapia Oncologica, A.O.U. San'T Orsola, Bologna
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale San Raffaele, Milan
  - Fondazione Policlinico Tor Vergata, Roma
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Azienda Ospedaliera Sant Andrea, Roma
- King Hussein Cancer Center, Amman, Jordan
- Lebanon (4):
  - St Georges Hospital university medical centre, Beirut
  - American Universitty of Beirut Medical Center, Beirut
  - Notre Dame De Secours, Byblos
  - Centre Hospitalier du Nord, Zghartā
- Mexico (7):
  - Consultorio de Especialidad en Urologia Privado, Durango
  - Hospital MAC Leon, León
  - Avix Investigacion Clinica S C, Monterrey
  - Oncologia Integral Satelite, Naucalpan
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
  - Oncocenter, Puebla City
  - Cuidados Oncologicos, Querétaro
- Poland (9):
  - Centrum Onkologii im Prof F Lukaszczyka w Bydgoszczy, Bydgoszcz
  - NU-MED Grupa S.A Centrum Radioterapii i Onkologii, Elblag
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpitale Pomorskie Sp z o o, Gdynia
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce
  - Szpital Wojewodzki im Mikolaja Kopernika w Koszalinie, Koszalin
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im M Kopernika w Lodzi, Lodz
  - Radomskie Centrum Onkologii, Radom
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Portugal (8):
  - Ipo Lisboa, Lisbon
  - Hosp. Cuf Tejo, Lisbon
  - Fund. Champalimaud, Lisbon
  - Uls Lisboa Ocidental - Hosp. Sao Francisco Xavier, Lisbon
  - Hosp. Da Luz Lisboa, Lisbon
  - Uls Santa Maria - Hosp. Santa Maria, Lisbon
  - Uls Santo Antonio - Hosp. Santo Antonio, Porto
  - Uls de Entre Douro E Vouga - Hosp. Sao Sebastiao, Santa Maria da Feira
- Russia (8):
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - City Clinical Hospital #57, Moscow
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - Hertzen Oncology Research Institute, Moscow
  - Leningrad Regional Oncology Dispensary, Saint Petersburg
  - SPb SBIH 'City Clinical Oncological Dispensary', Saint Petersburg
  - Multifunctional clinical medical center 'Medical city', Tyumen
  - SHI Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Slovakia (7):
  - CUIMED - urologická ambulancia, Bratislava
  - Východoslovenský Onkologický Ústav, Košice
  - Univerzitná nemocnica Martin, Martin
  - Uroexam s.r.o., Nitra
  - Urologicka ambulancia e.cho Poprad, s.r.o, Poprad
  - MILAB s.r.o., Prešov
  - Privátna urologická ambulancia, Trenčín
- Spain (11):
  - Hospital Universitario Puerto Del Mar, Cadiz
  - Hosp. Arquitecto Marcide, Ferrol
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. de La Paz, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. de Navarra, Pamplona
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. Clinico Univ. Lozano Blesa, Zaragoza
- Sweden (3):
  - Urologiska Mottagningen, Malmo
  - Prostatacancercentrum, Stockholm
  - Sodersjukhuset, Stockholm
- Turkey (Türkiye) (12):
  - Adana Baskent Yuregir Hospital, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Ankara University Medical Faculty, Ankara
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Koc University, School of Medicine, Koc University Hospital, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Bakirkoy Training and Research Hospital, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Kartal Dr Lutfi Kirdar Egitim ve Arastirma Hastanesi, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Sakarya Üniversitesi Tıp Fakültesi Hastanesi, Sakarya

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency